CLINICAL TRIAL: NCT02010658
Title: Effect of Cognitive Aid on Adherence to Perioperative Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Brigham and Women's Hospital (Other); University of Kentucky (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Model: Crossover | Purpose: Other
Other Study IDs: Pro00018749
Record Dates: First submitted 2013-12-01; First posted 2013-12-13 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Perioperative Decision Making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory (No Intervention)
- Cognitive Aid (Experimental)
  Interventions: Other: Cognitive Aid

INTERVENTIONS:
Other: Cognitive Aid
  Arms: Cognitive Aid

SUMMARY:
The objective of this prospective randomized trial is to ascertain whether the use of a cognitive aid improves adherence to best published practices for the management of simulated patients regarding perioperative cardiac evaluation and management.

ELIGIBILITY:
Inclusion Criteria:

Any active resident or faculty member will be allowed to volunteer.

Exclusion Criteria:

There are no exclusion criteria (notably we will include residents on academic probation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Adherence of ACC/AHA Guideline | Up to 6 weeks
  Adherence in terms of selection of the correct option for multiple choice question.

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Reeves, MD, Study Chair — Medical University of South Carolina